CLINICAL TRIAL: NCT01125124
Title: Evaluation of Chest Pain, Effectiveness and Safety of Pleurodesis With Pleural Catheters and Silver Nitrate for Malignant Pleural Effusion.
Brief Title: Safety and Effectiveness Study for Pleurodesis With Silver Nitrate in Malignant Pleural Effusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Dr Ricardo Mingarini Terra, INCOR-HCFMUSP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1041/09; 1041/09 (Other: University of Sao Paulo General Hospital Research Committee)
Record Dates: First submitted 2010-04-26; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Malignant Pleural Effusion
Keywords: Pleurodesis; Malignant pleural effusion; Silver Nitrate; Pain
MeSH Terms: conditions — Pleural Effusion, Malignant; Pain | interventions — Silver Nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Silver Nitrate 1 (Active Comparator): Patients submitted to pleurodesis via pleural catheter using 30ml of 0.5% silver nitrate solution.
  Interventions: Drug: Silver Nitrate
- Silver Nitrate 2 (Experimental): Patients submitted to instilation of 30ml 0.3% silver nitrate solution via pleural catheter.
  Interventions: Drug: Silver Nitrate
- Silver Nitrate 3 (Experimental): Patients submitted to instilation of 60ml 0.3% silver nitrate solution via pleural catheter.
  Interventions: Drug: Silver Nitrate

INTERVENTIONS:
Drug: Silver Nitrate — Instilation of silver nitrate solution through the pleural catheter. The catheter remains closed for 1h after the procedure and is then reopened. There will be 3 different dosages, corresponding to the 3 different arms.

SUMMARY:
The primary purpose of this study is to determinate the degree of chest pain on patients with malignant pleural effusion submitted to pleurodesis with silver nitrate in three different dosages and concentrations ( 30ml 0.5% ; 30ml 0.3% ; 60ml 0.3%). Our secondary purpose is to evaluate the efficacy and occurence of adverse effects in the usage of silver nitrate for pleurodesis in the aforementioned dosages/concentrations.

DETAILED DESCRIPTION:
Malignant pleural effusion is a frequent complication in advanced neoplasia. Pleurodesis is the procedure of choice for symptomatic control, with talc as the sclerosing agent of choice. However, the occurrence of severe adverse effects associated with its use has led to the search for other agents.

Silver nitrate poses an option, presenting excellent results in animal models and having successful usage in pleurodesis in the past. Although important, the current literature on the effective use of silver nitrate for pleurodesis is still too scarce, and a deeper knowledge on the occurrence of adverse side effects, especially pain, is still necessary to allow the substance to be considered as an effective alternative to talc, as well as for the definition of an adequate dosage.

ELIGIBILITY:
Inclusion Criteria:

* Malignant pleural effusion confirmed by cytologic analysis of the fluid and/or pleural biopsy.
* Recurrent and symptomatic malignant pleural effusion.
* Full pulmonary expansion (>90%) post thoracocentesis, confirmed via chest x-ray.
* Karnofsky Performance Status >30
* Agreement to participate of the study by signing of the Informed Consent Term.

Exclusion Criteria:

* Coagulopathies (prothrombin activity <50%) and/or thrombocytopenia (<80000 count).
* Active pleural or systemic infection.
* Massive skin neoplastic infiltration.
* Inability of understanding the pain scale.
* Previous pleural procedures (except for thoracocentesis and/or pleural biopsy).
* Refusal to participate of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Chest pain on the first five days after pleurodesis | Along the first five days after treatment
  Chest pain will be evaluated via Visual Analog Scale.
Chest pain after 10 days of pleurodesis | On the 10th day after the procedure.
  Chest pain will be assessed using the Visual Analog Scale
Chest pain after 30 days of pleurodesis | Within 30 days of the procedure
  Chest pain will be evaluated by Visual Analog Scale

SECONDARY OUTCOMES:
Effectiveness of the pleurodesis | After 30 days of the procedure
  On hospital discharge, five days after the procedure, patients are submitted to chest computerized tomography (CT). After 30 days of the procedure, patients are submitted to another chest CT and the volume of pleural effusion is calculated and compared to that of the hospital discharge date (calculated by the 5th day CT).
Dyspnea | Before the procedure, during the first five days after the procedure, ten days after the procedure and on the 30th day post-procedure.
  Dyspnea will be evaluated through the British MRC dyspnea scale.
Adverse effects | Within the first 5 days after the procedure, on the 10th day after the procedure and on the 30th day after the procedure
  The safety of the treatment will be assessed both by monitoring of complete blood counts, renal function, liver function and inflammation markers, as well as monitoring of body temperature, arterial blood pressure and heart rate. The occurrence of adverse side effects will be assessed using the United States National Cancer Institute Common Terminology Criteria for Adverse Events v.3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo M Terra, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Paschoalini Mda S, Vargas FS, Marchi E, Pereira JR, Jatene FB, Antonangelo L, Light RW. Prospective randomized trial of silver nitrate vs talc slurry in pleurodesis for symptomatic malignant pleural effusions. Chest. 2005 Aug;128(2):684-9. doi: 10.1378/chest.128.2.684. PMID 16100154